CLINICAL TRIAL: NCT04073940
Title: Exploration of Brain Changes Due to a Targeted Ballet Program in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Citlali Lopez-Ortiz, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18210
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; ataxia; magnetic resonance imaging; structural connectivity; resting state functional connectivity; dance; wellness; balance; mobility
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Ballet Program (Experimental): A 16-week (32 sessions of 1 hour each) ballet-based intervention targeted to improve motor function in persons with multiple sclerosis.
  Interventions: Behavioral: Targeted Ballet Program

INTERVENTIONS:
Behavioral: Targeted Ballet Program — All classes will be offered in a set schedule convenient for all participants. Classes will be taught by the PI, who has extensive dance training expertise. The targeted ballet program consists of an initial period of dance movements while sitting in chairs (20min), followed by exercises holding onto the ballet barres mounted to the walls in the Neuroscience of Dance on Health and Disability Laboratory (20min), followed by locomotive dance movements (20min). The dance moves are based on the Ballet I Syllabus of the Royal Academy of Dancing and the Cecchetti Council of America, designed for eight-year-old students with no necessary previous training in ballet.

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune disease of the central nervous system (CNS) affecting roughly 900,000 people in the United States that frequently results in impaired mobility. The majority of people with MS express that impaired mobility the most difficult aspect of living with the disease. Ataxia is one aspect of impaired mobility experienced by approximately 80% of persons with MS. Despite $9 billion in drug costs to patients with MS in the U.S., in 2012 alone, standard pharmacological treatment for MS is ineffective in restoring mobility and decreasing ataxia. The PI designed a targeted ballet program requiring motor learning of complex movements that mitigated ataxia and improved balance in patients with MS in a pilot study. The improvements obtained were approximately five times larger than those reported by other physical rehabilitation interventions. However, understanding these changes requires determining whether there are underlying changes in the brain after participation in the targeted ballet program.

This project involves persons with mild-to-moderate MS that present ataxia in their movement. We will compare the brain connectivity of participants in the targeted ballet program before and after the 16-week, twice per week, hourly participation intervention. Brain images will be obtained with magnetic resonance imaging while each participant rests with the eyes open. As a secondary outcome, measures of movement quality, ataxia, and balance will be taken to better understand the effects of the targeted ballet program on motor function, wellness, and the brains of persons with mild to moderate MS. Test on movement will include a 10 meter walk with motion tracking, a balance test using a force plate, and clinical tests of ataxia, balance, and walking speed. We will also assess changes in wellness with standard questionnaires.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune-mediated disease with brain demyelination and axonal loss that result in impaired mobility, which affects an estimated 75% of people with MS and is reported as the most difficult aspect of living with MS. An estimated 900,000 people in the U.S. suffer from MS, which has no known cure. In 2012 alone, drug costs to patients with MS in the U.S. were $9 billion. Despite the high costs, pharmacological interventions do not induce myelination so motor impairments persist. The PI designed a ballet-based program for complex motor learning delivered in a group setting. Our previous work provides evidence that the targeted ballet program increased balance and walking scores by 42% and decreased clinical ataxia scores by 58% over a period of 16 weeks and 32 hours of instruction. However, understanding these changes requires determining whether there are underlying changes in the brain after participation in the targeted ballet program.

The goal of this proposal is to provide evidence of improvements in brain connectivity measures after participation in the targeted ballet program in persons with MS. As secondary outcomes, we will assess motor function and wellness after participation in the targeted ballet program in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64
* Informed consent obtained
* Confirmation of relapsing remitting MS (RRMS) diagnosis by the participant's neurologist
* Presence of ataxia determined by the International Cooperative Ataxia Rating Scale (ICARS) recommended by the NIH and the Ataxia Neuropharmacology Committee of the World Federation of Neurology with a score greater or equal to 7
* Expanded Disability Status Scale (EDSS) scores of 1.0-6.5 based on an examination by a Neurostatus certified examiner for indicating walking impairment
* Relapse free in the previous 30 days
* Approval for exercise training.

Exclusion Criteria:

* Presence of severe cognitive impairment based on an oral Symbol Digit Modalities Test (SDMT) score of less than 23, or the Montreal Cognitive Assessment (MoCA) Test less than 22
* Inability to understand experimental instructions presented in English
* Pregnancy
* Education level less than 8th grade - due to concerns about understanding the study and consent form
* Change in use of disease modifying therapy in the previous 6 months,
* Initiation of Ampyra or other medications that influence walking and mobility within the previous 30 days,
* History of brain injury or central nervous system disease other than multiple sclerosis - this will be determined from gross anatomical abnormalities in the images or from medical history on Biomedical Imaging Center (BIC) screening form,
* Presence of orthopedic conditions,
* The presence of any skin conditions preventing the safe usage of motion tracking marker adhesives
* The presence of conditions which would contra-indicate MRI: prior surgeries and/or implant of pacemakers, pacemaker wires, artificial heart valve, brain aneurysm surgery, middle ear implant, non-removable hearing aid or jewelry, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, artificial limb or joint; foreign metallic objects in the body such as bullets, BB's, shrapnel, or metalwork fragments; pregnancy, claustrophobia, uncontrollable shaking, or inability to lie still for 2 hours.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Structural Connectivity | Before and after the 16-week intervention period
  Mean strength, global efficiency, and mean clustering coefficient for the networks seeded from the regions of interest: the fornix, supplemental motor area, corpus callosum, orbitofrontal cortex, putamen, and cerebellum. Using Probtrackx2 in network mode, the output is a connectivity martix, which contains the number of streamlines from each seed volume (e.g., all voxels in insula cortex) that reached all other target regions. Structural connections will be normalized by the average volume of each region of interest (ROI) comprising the particular pathway to eliminate bias induced from larger ROI's. Additionally, the structural connectomes will be symmetrized by averaging the two connections in the connectivity matrix corresponding to the pair of ROI's (where one connection is ROI 1 as seed and ROI 2 as target, and the other connection flips the seed and target labels).
Resting-State Functional Connectivity | Before and after the 16-week intervention period
  We will acquire one 8 minute scan for resting state functional connectivity analysis, during which participants will be instructed to maintain their eyes open and focus on a fixation point as was done in Bollaert et al. 2018. We will use a modified version of the Duke Brain Imaging and Analysis Center's (BIAC) resting-state functional connectivity to find the correlation coefficients of the resting-state blood oxygen level-dependent activation of the 68 regions from Freesurfer's parcellation and the 34 regions of the cerebellum from the spatially unbiased atlas template of the cerebellum and brainstem (SUIT) parcellation. We will use the brain connectivity toolbox (BCT) to form graph-theoretical measures of the network for evaluating changes in connectivity.

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale (ICARS) | Before and after the 16-week intervention period
  The ICARS is the leading comprehensive clinical measure of ataxia for persons with MS, which has strong inter-evaluator reliability and validity.
Mini Balance Evaluation Systems Test (Mini-BESTest) | Before and after the 16-week intervention period
  This test consists of a shorter list of evaluations on six factors that may impair balance in patients with MS: biomechanics, stability limits, postural responses, anticipatory postural adjustments, sensory orientation, and dynamic balance during gait.
10-Meter Walk Test (10MWT) | Before and after the 16-week intervention period
  A clinical test of walking ability by time to complete a 10-meter long walk.
World Health Organization Disability Assessment Schedule (WHODAS) | Before and after the 16-week intervention period
  Questionnaire-based assessment of wellness and quality of life as related to disability. 36 items are used to assess disability-related wellness. Difficulty in the past 30 days for each item is scored between 1 (none) and 5 (extreme or cannot do). Six domains are assessed: Understanding and communicating (6 to 30), Getting around (5 to 25), Self-care (4 to 20), Getting along with people (5 to 25), Life activities (8 to 40), and Participation in society (8 to 40) The minimum sum score of 36 indicates no disability-related wellness problems and the maximum score of 180 indicates extreme disability-related wellness problems.
World Health Organization Five Well-Being Index (WHO-5). | Before and after the 16-week intervention period
  Questionnaire-based assessment of wellness and quality of life over the last two weeks. A minimum sum score of 0 (0 on each of five questions) indicates minimal well-being. A maximum score of 25 (5 on each of five questions) indicates maximum well-being.
Smoothness Index | Before and after the 16-week intervention period
  Quantitative measure of smoothness of movement will be obtained for walking by computing a standard smoothness index on velocity data of body landmarks such as wrists, elbows, shoulders, hips, knees, toes, ankles, and top of head in a 5 meter walk using a motion capture system (Qualisys, Sweden).
Step-to-Stand Stabilization Task | Before and after the 16-week intervention period
  Participant will step onto and stand still on a force plate to quantitatively measure static and dynamic balance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data will be kept for 5 years after publication, as required by the American Psychological Association. De-identified data will be stored in the Neuroscience Information Framework database for further use.

REFERENCES:
- [Background] Bollaert RE, Poe K, Hubbard EA, Motl RW, Pilutti LA, Johnson CL, Sutton BP. Associations of functional connectivity and walking performance in multiple sclerosis. Neuropsychologia. 2018 Aug;117:8-12. doi: 10.1016/j.neuropsychologia.2018.05.007. Epub 2018 May 8. PMID 29750986
- [Background] Scheidler AM, Kinnett-Hopkins D, Learmonth YC, Motl R, Lopez-Ortiz C. Targeted ballet program mitigates ataxia and improves balance in females with mild-to-moderate multiple sclerosis. PLoS One. 2018 Oct 18;13(10):e0205382. doi: 10.1371/journal.pone.0205382. eCollection 2018. PMID 30335774
- [Background] Larocca NG. Impact of walking impairment in multiple sclerosis: perspectives of patients and care partners. Patient. 2011;4(3):189-201. doi: 10.2165/11591150-000000000-00000. PMID 21766914
- [Background] Mills RJ, Yap L, Young CA. Treatment for ataxia in multiple sclerosis. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD005029. doi: 10.1002/14651858.CD005029.pub2. PMID 17253537
- [Background] Wallin MT, Culpepper WJ, Campbell JD, Nelson LM, Langer-Gould A, Marrie RA, Cutter GR, Kaye WE, Wagner L, Tremlett H, Buka SL, Dilokthornsakul P, Topol B, Chen LH, LaRocca NG; US Multiple Sclerosis Prevalence Workgroup. The prevalence of MS in the United States: A population-based estimate using health claims data. Neurology. 2019 Mar 5;92(10):e1029-e1040. doi: 10.1212/WNL.0000000000007035. Epub 2019 Feb 15. PMID 30770430
- [Background] Hartung DM, Bourdette DN, Ahmed SM, Whitham RH. The cost of multiple sclerosis drugs in the US and the pharmaceutical industry: Too big to fail? Neurology. 2015 May 26;84(21):2185-92. doi: 10.1212/WNL.0000000000001608. Epub 2015 Apr 24. PMID 25911108
- [Background] Lakhani B, Borich MR, Jackson JN, Wadden KP, Peters S, Villamayor A, MacKay AL, Vavasour IM, Rauscher A, Boyd LA. Motor Skill Acquisition Promotes Human Brain Myelin Plasticity. Neural Plast. 2016;2016:7526135. doi: 10.1155/2016/7526135. Epub 2016 May 16. PMID 27293906
- [Background] Wittenberg GF, Richards LG, Jones-Lush LM, Roys SR, Gullapalli RP, Yang S, Guarino PD, Lo AC. Predictors and brain connectivity changes associated with arm motor function improvement from intensive practice in chronic stroke. F1000Res. 2016 Aug 31;5:2119. doi: 10.12688/f1000research.8603.2. eCollection 2016. PMID 28357039
- [Background] Solesio-Jofre E, Beets IAM, Woolley DG, Pauwels L, Chalavi S, Mantini D, Swinnen SP. Age-Dependent Modulations of Resting State Connectivity Following Motor Practice. Front Aging Neurosci. 2018 Feb 6;10:25. doi: 10.3389/fnagi.2018.00025. eCollection 2018. PMID 29467646
- [Background] Scholz J, Klein MC, Behrens TE, Johansen-Berg H. Training induces changes in white-matter architecture. Nat Neurosci. 2009 Nov;12(11):1370-1. doi: 10.1038/nn.2412. Epub 2009 Oct 11. PMID 19820707
- [Background] Taubert M, Draganski B, Anwander A, Muller K, Horstmann A, Villringer A, Ragert P. Dynamic properties of human brain structure: learning-related changes in cortical areas and associated fiber connections. J Neurosci. 2010 Sep 1;30(35):11670-7. doi: 10.1523/JNEUROSCI.2567-10.2010. PMID 20810887
- [Background] Moore E, Schaefer RS, Bastin ME, Roberts N, Overy K. Diffusion tensor MRI tractography reveals increased fractional anisotropy (FA) in arcuate fasciculus following music-cued motor training. Brain Cogn. 2017 Aug;116:40-46. doi: 10.1016/j.bandc.2017.05.001. Epub 2017 Jun 12. PMID 28618361
- [Background] Burzynska AZ, Jiao Y, Knecht AM, Fanning J, Awick EA, Chen T, Gothe N, Voss MW, McAuley E, Kramer AF. White Matter Integrity Declined Over 6-Months, but Dance Intervention Improved Integrity of the Fornix of Older Adults. Front Aging Neurosci. 2017 Mar 16;9:59. doi: 10.3389/fnagi.2017.00059. eCollection 2017. PMID 28360853
- [Background] Clayden JD. Imaging connectivity: MRI and the structural networks of the brain. Funct Neurol. 2013 Jul-Sep;28(3):197-203. PMID 24139656
- [Background] Beaulieu C. The basis of anisotropic water diffusion in the nervous system - a technical review. NMR Biomed. 2002 Nov-Dec;15(7-8):435-55. doi: 10.1002/nbm.782. PMID 12489094
- [Background] Seehaus A, Roebroeck A, Bastiani M, Fonseca L, Bratzke H, Lori N, Vilanova A, Goebel R, Galuske R. Histological validation of high-resolution DTI in human post mortem tissue. Front Neuroanat. 2015 Jul 23;9:98. doi: 10.3389/fnana.2015.00098. eCollection 2015. PMID 26257612
- [Background] Friston KJ. Functional and effective connectivity: a review. Brain Connect. 2011;1(1):13-36. doi: 10.1089/brain.2011.0008. PMID 22432952
- [Background] Brunberg JA; Expert Panel on Neurologic Imaging. Ataxia. AJNR Am J Neuroradiol. 2008 Aug;29(7):1420-2. No abstract available. PMID 18701585
- [Background] Vargas DL, Tyor WR. Update on disease-modifying therapies for multiple sclerosis. J Investig Med. 2017 Jun;65(5):883-891. doi: 10.1136/jim-2016-000339. Epub 2017 Jan 27. PMID 28130412
- [Background] Akaishi T, Nakashima I. Efficiency of antibody therapy in demyelinating diseases. Int Immunol. 2017 Jul 1;29(7):327-335. doi: 10.1093/intimm/dxx037. PMID 28910968
- [Background] Sternad D, Marino H, Charles SK, Duarte M, Dipietro L, Hogan N. Transitions between discrete and rhythmic primitives in a unimanual task. Front Comput Neurosci. 2013 Jul 22;7:90. doi: 10.3389/fncom.2013.00090. eCollection 2013. PMID 23888139
- [Background] Flash T, Hogan N. The coordination of arm movements: an experimentally confirmed mathematical model. J Neurosci. 1985 Jul;5(7):1688-703. doi: 10.1523/JNEUROSCI.05-07-01688.1985. PMID 4020415
- [Background] Lopez-Ortiz C, Gaebler-Spira DJ, Mckeeman SN, Mcnish RN, Green D. Dance and rehabilitation in cerebral palsy: a systematic search and review. Dev Med Child Neurol. 2019 Apr;61(4):393-398. doi: 10.1111/dmcn.14064. Epub 2018 Oct 23. PMID 30350851
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Kraft GH. Rehabilitation still the only way to improve function in multiple sclerosis. Lancet. 1999 Dec 11;354(9195):2016-7. doi: 10.1016/S0140-6736(99)90035-1. No abstract available. PMID 10636362
- [Background] Gosney JL, Scott JA, Snook EM, Motl RW. Physical activity and multiple sclerosis: validity of self-report and objective measures. Fam Community Health. 2007 Apr-Jun;30(2):144-50. doi: 10.1097/01.fch.0000264411.20766.0c. PMID 19241650
- [Background] Snook EM, Motl RW. Effect of exercise training on walking mobility in multiple sclerosis: a meta-analysis. Neurorehabil Neural Repair. 2009 Feb;23(2):108-16. doi: 10.1177/1545968308320641. Epub 2008 Oct 23. PMID 18948413
- [Background] Tarakci E, Yeldan I, Huseyinsinoglu BE, Zenginler Y, Eraksoy M. Group exercise training for balance, functional status, spasticity, fatigue and quality of life in multiple sclerosis: a randomized controlled trial. Clin Rehabil. 2013 Sep;27(9):813-22. doi: 10.1177/0269215513481047. Epub 2013 Mar 29. PMID 23543341
- [Background] Gunn H, Markevics S, Haas B, Marsden J, Freeman J. Systematic Review: The Effectiveness of Interventions to Reduce Falls and Improve Balance in Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2015 Oct;96(10):1898-912. doi: 10.1016/j.apmr.2015.05.018. Epub 2015 Jun 10. PMID 26070975
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890
- [Background] Mandelbaum R, Triche EW, Fasoli SE, Lo AC. A Pilot Study: examining the effects and tolerability of structured dance intervention for individuals with multiple sclerosis. Disabil Rehabil. 2016;38(3):218-22. doi: 10.3109/09638288.2015.1035457. Epub 2015 Apr 15. PMID 25875049
- [Background] Kiefer AW, Riley MA, Shockley K, Sitton CA, Hewett TE, Cummins-Sebree S, Haas JG. Lower-limb proprioceptive awareness in professional ballet dancers. J Dance Med Sci. 2013 Sep;17(3):126-32. doi: 10.12678/1089-313x.17.3.126. PMID 24069947
- [Background] Schmit JM, Regis DI, Riley MA. Dynamic patterns of postural sway in ballet dancers and track athletes. Exp Brain Res. 2005 Jun;163(3):370-8. doi: 10.1007/s00221-004-2185-6. Epub 2005 Jan 18. PMID 15655686
- [Background] Thullier F, Moufti H. Multi-joint coordination in ballet dancers. Neurosci Lett. 2004 Oct 7;369(1):80-4. doi: 10.1016/j.neulet.2004.08.011. PMID 15380312
- [Background] Lepelley MC, Thullier F, Koral J, Lestienne FG. Muscle coordination in complex movements during Jete in skilled ballet dancers. Exp Brain Res. 2006 Nov;175(2):321-31. doi: 10.1007/s00221-006-0552-1. Epub 2006 Jun 2. PMID 16741715
- [Background] Jola C, Davis A, Haggard P. Proprioceptive integration and body representation: insights into dancers' expertise. Exp Brain Res. 2011 Sep;213(2-3):257-65. doi: 10.1007/s00221-011-2743-7. Epub 2011 Jun 4. PMID 21643713
- [Background] Ramsay JR, Riddoch MJ. Position-matching in the upper limb: professional ballet dancers perform with outstanding accuracy. Clin Rehabil. 2001 Jun;15(3):324-30. doi: 10.1191/026921501666288152. PMID 11386404
- [Background] Hanggi J, Koeneke S, Bezzola L, Jancke L. Structural neuroplasticity in the sensorimotor network of professional female ballet dancers. Hum Brain Mapp. 2010 Aug;31(8):1196-206. doi: 10.1002/hbm.20928. PMID 20024944
- [Background] Ng A, Bunyan S, Suh J, Huenink P, Gregory T, Gambon S, Miller D. Ballroom dance for persons with multiple sclerosis: a pilot feasibility study. Disabil Rehabil. 2020 Apr;42(8):1115-1121. doi: 10.1080/09638288.2018.1516817. Epub 2019 Jan 13. PMID 30638081
- [Background] McKenzie IA, Ohayon D, Li H, de Faria JP, Emery B, Tohyama K, Richardson WD. Motor skill learning requires active central myelination. Science. 2014 Oct 17;346(6207):318-22. doi: 10.1126/science.1254960. PMID 25324381
- [Background] Gibson EM, Purger D, Mount CW, Goldstein AK, Lin GL, Wood LS, Inema I, Miller SE, Bieri G, Zuchero JB, Barres BA, Woo PJ, Vogel H, Monje M. Neuronal activity promotes oligodendrogenesis and adaptive myelination in the mammalian brain. Science. 2014 May 2;344(6183):1252304. doi: 10.1126/science.1252304. Epub 2014 Apr 10. PMID 24727982
- [Background] Chang EH, Argyelan M, Aggarwal M, Chandon TS, Karlsgodt KH, Mori S, Malhotra AK. The role of myelination in measures of white matter integrity: Combination of diffusion tensor imaging and two-photon microscopy of CLARITY intact brains. Neuroimage. 2017 Feb 15;147:253-261. doi: 10.1016/j.neuroimage.2016.11.068. Epub 2016 Dec 13. PMID 27986605
- [Background] Laule C, Leung E, Lis DK, Traboulsee AL, Paty DW, MacKay AL, Moore GR. Myelin water imaging in multiple sclerosis: quantitative correlations with histopathology. Mult Scler. 2006 Dec;12(6):747-53. doi: 10.1177/1352458506070928. PMID 17263002
- [Background] Baer LH, Park MT, Bailey JA, Chakravarty MM, Li KZ, Penhune VB. Regional cerebellar volumes are related to early musical training and finger tapping performance. Neuroimage. 2015 Apr 1;109:130-9. doi: 10.1016/j.neuroimage.2014.12.076. Epub 2015 Jan 9. PMID 25583606
- [Background] Biswal BB, Mennes M, Zuo XN, Gohel S, Kelly C, Smith SM, Beckmann CF, Adelstein JS, Buckner RL, Colcombe S, Dogonowski AM, Ernst M, Fair D, Hampson M, Hoptman MJ, Hyde JS, Kiviniemi VJ, Kotter R, Li SJ, Lin CP, Lowe MJ, Mackay C, Madden DJ, Madsen KH, Margulies DS, Mayberg HS, McMahon K, Monk CS, Mostofsky SH, Nagel BJ, Pekar JJ, Peltier SJ, Petersen SE, Riedl V, Rombouts SA, Rypma B, Schlaggar BL, Schmidt S, Seidler RD, Siegle GJ, Sorg C, Teng GJ, Veijola J, Villringer A, Walter M, Wang L, Weng XC, Whitfield-Gabrieli S, Williamson P, Windischberger C, Zang YF, Zhang HY, Castellanos FX, Milham MP. Toward discovery science of human brain function. Proc Natl Acad Sci U S A. 2010 Mar 9;107(10):4734-9. doi: 10.1073/pnas.0911855107. Epub 2010 Feb 22. PMID 20176931
- [Background] Leavitt VM, Cirnigliaro C, Cohen A, Farag A, Brooks M, Wecht JM, Wylie GR, Chiaravalloti ND, DeLuca J, Sumowski JF. Aerobic exercise increases hippocampal volume and improves memory in multiple sclerosis: preliminary findings. Neurocase. 2014;20(6):695-7. doi: 10.1080/13554794.2013.841951. Epub 2013 Oct 4. PMID 24090098
- [Background] Pinter D, Beckmann C, Koini M, Pirker E, Filippini N, Pichler A, Fuchs S, Fazekas F, Enzinger C. Reproducibility of Resting State Connectivity in Patients with Stable Multiple Sclerosis. PLoS One. 2016 Mar 23;11(3):e0152158. doi: 10.1371/journal.pone.0152158. eCollection 2016. PMID 27007237
- [Background] Rocca MA, Valsasina P, Leavitt VM, Rodegher M, Radaelli M, Riccitelli GC, Martinelli V, Martinelli-Boneschi F, Falini A, Comi G, Filippi M. Functional network connectivity abnormalities in multiple sclerosis: Correlations with disability and cognitive impairment. Mult Scler. 2018 Apr;24(4):459-471. doi: 10.1177/1352458517699875. Epub 2017 Mar 15. PMID 28294693
- [Background] Dogonowski AM, Andersen KW, Madsen KH, Sorensen PS, Paulson OB, Blinkenberg M, Siebner HR. Multiple sclerosis impairs regional functional connectivity in the cerebellum. Neuroimage Clin. 2013 Nov 27;4:130-8. doi: 10.1016/j.nicl.2013.11.005. eCollection 2014. PMID 24371795
- [Background] Demirakca T, Cardinale V, Dehn S, Ruf M, Ende G. The Exercising Brain: Changes in Functional Connectivity Induced by an Integrated Multimodal Cognitive and Whole-Body Coordination Training. Neural Plast. 2016;2016:8240894. doi: 10.1155/2016/8240894. Epub 2015 Dec 27. PMID 26819776
- [Background] Sandroff BM, Wylie GR, Sutton BP, Johnson CL, DeLuca J, Motl RW. Treadmill walking exercise training and brain function in multiple sclerosis: Preliminary evidence setting the stage for a network-based approach to rehabilitation. Mult Scler J Exp Transl Clin. 2018 Feb 21;4(1):2055217318760641. doi: 10.1177/2055217318760641. eCollection 2018 Jan-Mar. PMID 29497559
- [Background] McGregor HR, Gribble PL. Changes in visual and sensory-motor resting-state functional connectivity support motor learning by observing. J Neurophysiol. 2015 Jul;114(1):677-88. doi: 10.1152/jn.00286.2015. Epub 2015 May 20. PMID 25995349
- [Background] McGregor HR, Cashaback JGA, Gribble PL. Somatosensory perceptual training enhances motor learning by observing. J Neurophysiol. 2018 Dec 1;120(6):3017-3025. doi: 10.1152/jn.00313.2018. Epub 2018 Sep 19. PMID 30230990
- [Background] Grebenciucova E, Pruitt A. Infections in Patients Receiving Multiple Sclerosis Disease-Modifying Therapies. Curr Neurol Neurosci Rep. 2017 Sep 22;17(11):88. doi: 10.1007/s11910-017-0800-8. PMID 28940162
- [Background] Sampaio-Baptista C, Khrapitchev AA, Foxley S, Schlagheck T, Scholz J, Jbabdi S, DeLuca GC, Miller KL, Taylor A, Thomas N, Kleim J, Sibson NR, Bannerman D, Johansen-Berg H. Motor skill learning induces changes in white matter microstructure and myelination. J Neurosci. 2013 Dec 11;33(50):19499-503. doi: 10.1523/JNEUROSCI.3048-13.2013. PMID 24336716
- [Background] Barclay A, Paul L, MacFarlane N, McFadyen AK. The effect of cycling using active-passive trainers on spasticity, cardiovascular fitness, function and quality of life in people with moderate to severe Multiple Sclerosis (MS); a feasibility study. Mult Scler Relat Disord. 2019 Sep;34:128-134. doi: 10.1016/j.msard.2019.06.019. Epub 2019 Jun 18. PMID 31260943
- [Background] Sadeghi Bahmani D, Kesselring J, Papadimitriou M, Bansi J, Puhse U, Gerber M, Shaygannejad V, Holsboer-Trachsler E, Brand S. In Patients With Multiple Sclerosis, Both Objective and Subjective Sleep, Depression, Fatigue, and Paresthesia Improved After 3 Weeks of Regular Exercise. Front Psychiatry. 2019 May 3;10:265. doi: 10.3389/fpsyt.2019.00265. eCollection 2019. PMID 31130879
- [Background] Hoff M, Kaminski E, Rjosk V, Sehm B, Steele CJ, Villringer A, Ragert P. Augmenting mirror visual feedback-induced performance improvements in older adults. Eur J Neurosci. 2015 May;41(11):1475-83. doi: 10.1111/ejn.12899. Epub 2015 Apr 24. PMID 25912048
- [Background] Storey E, Tuck K, Hester R, Hughes A, Churchyard A. Inter-rater reliability of the International Cooperative Ataxia Rating Scale (ICARS). Mov Disord. 2004 Feb;19(2):190-2. doi: 10.1002/mds.10657. PMID 14978674
- [Background] Trouillas P, Takayanagi T, Hallett M, Currier RD, Subramony SH, Wessel K, Bryer A, Diener HC, Massaquoi S, Gomez CM, Coutinho P, Ben Hamida M, Campanella G, Filla A, Schut L, Timann D, Honnorat J, Nighoghossian N, Manyam B. International Cooperative Ataxia Rating Scale for pharmacological assessment of the cerebellar syndrome. The Ataxia Neuropharmacology Committee of the World Federation of Neurology. J Neurol Sci. 1997 Feb 12;145(2):205-11. doi: 10.1016/s0022-510x(96)00231-6. PMID 9094050
- [Background] Salci Y, Fil A, Keklicek H, Cetin B, Armutlu K, Dolgun A, Tuncer A, Karabudak R. Validity and reliability of the International Cooperative Ataxia Rating Scale (ICARS) and the Scale for the Assessment and Rating of Ataxia (SARA) in multiple sclerosis patients with ataxia. Mult Scler Relat Disord. 2017 Nov;18:135-140. doi: 10.1016/j.msard.2017.09.032. Epub 2017 Sep 29. PMID 29141795
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] Potter K, Anderberg L, Anderson D, Bauer B, Beste M, Navrat S, Kohia M. Reliability, validity, and responsiveness of the Balance Evaluation Systems Test (BESTest) in individuals with multiple sclerosis. Physiotherapy. 2018 Mar;104(1):142-148. doi: 10.1016/j.physio.2017.06.001. Epub 2017 Jun 17. PMID 28888670
- [Background] Mitchell KD, Chen H, Silfies SP. Test-Retest Reliability, Validity, and Minimal Detectable Change of the Balance Evaluation Systems Test to Assess Balance in Persons with Multiple Sclerosis. Int J MS Care. 2018 Sep-Oct;20(5):231-237. doi: 10.7224/1537-2073.2016-118. PMID 30374253
- [Background] Balasubramanian S, Melendez-Calderon A, Burdet E. A robust and sensitive metric for quantifying movement smoothness. IEEE Trans Biomed Eng. 2012 Aug;59(8):2126-36. doi: 10.1109/TBME.2011.2179545. Epub 2011 Dec 13. PMID 22180502
- [Background] Gage WH, Winter DA, Frank JS, Adkin AL. Kinematic and kinetic validity of the inverted pendulum model in quiet standing. Gait Posture. 2004 Apr;19(2):124-32. doi: 10.1016/S0966-6362(03)00037-7. PMID 15013500
- [Background] Winter DA, Patla AE, Prince F, Ishac M, Gielo-Perczak K. Stiffness control of balance in quiet standing. J Neurophysiol. 1998 Sep;80(3):1211-21. doi: 10.1152/jn.1998.80.3.1211. PMID 9744933
- [Background] Altilio R, Paoloni M, Panella M. Selection of clinical features for pattern recognition applied to gait analysis. Med Biol Eng Comput. 2017 Apr;55(4):685-695. doi: 10.1007/s11517-016-1546-1. Epub 2016 Jul 19. PMID 27435068
- [Background] Givon U, Zeilig G, Achiron A. Gait analysis in multiple sclerosis: characterization of temporal-spatial parameters using GAITRite functional ambulation system. Gait Posture. 2009 Jan;29(1):138-42. doi: 10.1016/j.gaitpost.2008.07.011. Epub 2008 Oct 31. PMID 18951800
- [Background] Socie MJ, Motl RW, Pula JH, Sandroff BM, Sosnoff JJ. Gait variability and disability in multiple sclerosis. Gait Posture. 2013 May;38(1):51-5. doi: 10.1016/j.gaitpost.2012.10.012. Epub 2012 Nov 13. PMID 23153835
- [Background] Kalron A. Gait variability across the disability spectrum in people with multiple sclerosis. J Neurol Sci. 2016 Feb 15;361:1-6. doi: 10.1016/j.jns.2015.12.012. Epub 2015 Dec 10. PMID 26810506
- [Background] Auerbach EJ, Xu J, Yacoub E, Moeller S, Ugurbil K. Multiband accelerated spin-echo echo planar imaging with reduced peak RF power using time-shifted RF pulses. Magn Reson Med. 2013 May;69(5):1261-7. doi: 10.1002/mrm.24719. Epub 2013 Mar 6. PMID 23468087
- [Background] Setsompop K, Gagoski BA, Polimeni JR, Witzel T, Wedeen VJ, Wald LL. Blipped-controlled aliasing in parallel imaging for simultaneous multislice echo planar imaging with reduced g-factor penalty. Magn Reson Med. 2012 May;67(5):1210-24. doi: 10.1002/mrm.23097. Epub 2011 Aug 19. PMID 21858868
- [Background] Setsompop K, Cohen-Adad J, Gagoski BA, Raij T, Yendiki A, Keil B, Wedeen VJ, Wald LL. Improving diffusion MRI using simultaneous multi-slice echo planar imaging. Neuroimage. 2012 Oct 15;63(1):569-80. doi: 10.1016/j.neuroimage.2012.06.033. Epub 2012 Jun 23. PMID 22732564
- [Background] Xu J, Moeller S, Auerbach EJ, Strupp J, Smith SM, Feinberg DA, Yacoub E, Ugurbil K. Evaluation of slice accelerations using multiband echo planar imaging at 3 T. Neuroimage. 2013 Dec;83:991-1001. doi: 10.1016/j.neuroimage.2013.07.055. Epub 2013 Jul 27. PMID 23899722
- [Background] Wetter NC, Hubbard EA, Motl RW, Sutton BP. Fully automated open-source lesion mapping of T2-FLAIR images with FSL correlates with clinical disability in MS. Brain Behav. 2016 Jan 28;6(3):e00440. doi: 10.1002/brb3.440. eCollection 2016 Mar. PMID 26855828
- [Background] Davis SW, Dennis NA, Buchler NG, White LE, Madden DJ, Cabeza R. Assessing the effects of age on long white matter tracts using diffusion tensor tractography. Neuroimage. 2009 Jun;46(2):530-41. doi: 10.1016/j.neuroimage.2009.01.068. PMID 19385018
- [Background] Hubbard EA, Wetter NC, Sutton BP, Pilutti LA, Motl RW. Diffusion tensor imaging of the corticospinal tract and walking performance in multiple sclerosis. J Neurol Sci. 2016 Apr 15;363:225-31. doi: 10.1016/j.jns.2016.02.044. Epub 2016 Feb 18. PMID 27000254
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092
- [Background] Andersson JLR, Sotiropoulos SN. An integrated approach to correction for off-resonance effects and subject movement in diffusion MR imaging. Neuroimage. 2016 Jan 15;125:1063-1078. doi: 10.1016/j.neuroimage.2015.10.019. Epub 2015 Oct 20. PMID 26481672
- [Background] Smith SM, Jenkinson M, Johansen-Berg H, Rueckert D, Nichols TE, Mackay CE, Watkins KE, Ciccarelli O, Cader MZ, Matthews PM, Behrens TE. Tract-based spatial statistics: voxelwise analysis of multi-subject diffusion data. Neuroimage. 2006 Jul 15;31(4):1487-505. doi: 10.1016/j.neuroimage.2006.02.024. Epub 2006 Apr 19. PMID 16624579
- [Background] Winkler AM, Ridgway GR, Webster MA, Smith SM, Nichols TE. Permutation inference for the general linear model. Neuroimage. 2014 May 15;92(100):381-97. doi: 10.1016/j.neuroimage.2014.01.060. Epub 2014 Feb 11. PMID 24530839
- [Background] Smith SM, Nichols TE. Threshold-free cluster enhancement: addressing problems of smoothing, threshold dependence and localisation in cluster inference. Neuroimage. 2009 Jan 1;44(1):83-98. doi: 10.1016/j.neuroimage.2008.03.061. Epub 2008 Apr 11. PMID 18501637
- [Background] Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. Hum Brain Mapp. 1999;8(4):272-84. doi: 10.1002/(sici)1097-0193(1999)8:43.0.co;2-4. PMID 10619420
- [Background] Diedrichsen J, Zotow E. Surface-Based Display of Volume-Averaged Cerebellar Imaging Data. PLoS One. 2015 Jul 31;10(7):e0133402. doi: 10.1371/journal.pone.0133402. eCollection 2015. PMID 26230510
- [Background] Diedrichsen J, Maderwald S, Kuper M, Thurling M, Rabe K, Gizewski ER, Ladd ME, Timmann D. Imaging the deep cerebellar nuclei: a probabilistic atlas and normalization procedure. Neuroimage. 2011 Feb 1;54(3):1786-94. doi: 10.1016/j.neuroimage.2010.10.035. Epub 2010 Oct 18. PMID 20965257
- [Background] Diedrichsen J, Balsters JH, Flavell J, Cussans E, Ramnani N. A probabilistic MR atlas of the human cerebellum. Neuroimage. 2009 May 15;46(1):39-46. doi: 10.1016/j.neuroimage.2009.01.045. Epub 2009 Feb 5. PMID 19457380
- [Background] Diedrichsen J. A spatially unbiased atlas template of the human cerebellum. Neuroimage. 2006 Oct 15;33(1):127-38. doi: 10.1016/j.neuroimage.2006.05.056. Epub 2006 Aug 14. PMID 16904911
- [Background] Behrens TE, Berg HJ, Jbabdi S, Rushworth MF, Woolrich MW. Probabilistic diffusion tractography with multiple fibre orientations: What can we gain? Neuroimage. 2007 Jan 1;34(1):144-55. doi: 10.1016/j.neuroimage.2006.09.018. Epub 2006 Oct 27. PMID 17070705
- [Background] Sharp PB, Sutton BP, Paul EJ, Sherepa N, Hillman CH, Cohen NJ, Kramer AF, Prakash RS, Heller W, Telzer EH, Barbey AK. Mindfulness training induces structural connectome changes in insula networks. Sci Rep. 2018 May 21;8(1):7929. doi: 10.1038/s41598-018-26268-w. PMID 29785055
- [Background] Rubinov M, Sporns O. Complex network measures of brain connectivity: uses and interpretations. Neuroimage. 2010 Sep;52(3):1059-69. doi: 10.1016/j.neuroimage.2009.10.003. Epub 2009 Oct 9. PMID 19819337
- [Background] Chen NK, Chou YH, Song AW, Madden DJ. Measurement of spontaneous signal fluctuations in fMRI: adult age differences in intrinsic functional connectivity. Brain Struct Funct. 2009 Oct;213(6):571-85. doi: 10.1007/s00429-009-0218-4. Epub 2009 Sep 2. PMID 19727810
- [Background] Wakana S, Caprihan A, Panzenboeck MM, Fallon JH, Perry M, Gollub RL, Hua K, Zhang J, Jiang H, Dubey P, Blitz A, van Zijl P, Mori S. Reproducibility of quantitative tractography methods applied to cerebral white matter. Neuroimage. 2007 Jul 1;36(3):630-44. doi: 10.1016/j.neuroimage.2007.02.049. Epub 2007 Mar 20. PMID 17481925
- [Background] Hua K, Zhang J, Wakana S, Jiang H, Li X, Reich DS, Calabresi PA, Pekar JJ, van Zijl PC, Mori S. Tract probability maps in stereotaxic spaces: analyses of white matter anatomy and tract-specific quantification. Neuroimage. 2008 Jan 1;39(1):336-47. doi: 10.1016/j.neuroimage.2007.07.053. Epub 2007 Aug 15. PMID 17931890
- [Background] Guglielmetti C, Veraart J, Roelant E, Mai Z, Daans J, Van Audekerke J, Naeyaert M, Vanhoutte G, Delgado Y Palacios R, Praet J, Fieremans E, Ponsaerts P, Sijbers J, Van der Linden A, Verhoye M. Diffusion kurtosis imaging probes cortical alterations and white matter pathology following cuprizone induced demyelination and spontaneous remyelination. Neuroimage. 2016 Jan 15;125:363-377. doi: 10.1016/j.neuroimage.2015.10.052. Epub 2015 Oct 23. PMID 26525654
- [Background] Magistrale G, Pisani V, Argento O, Incerti CC, Bozzali M, Cadavid D, Caltagirone C, Medori R, DeLuca J, Nocentini U. Validation of the World Health Organization Disability Assessment Schedule II (WHODAS-II) in patients with multiple sclerosis. Mult Scler. 2015 Apr;21(4):448-56. doi: 10.1177/1352458514543732. Epub 2014 Aug 4. PMID 25092769
- [Background] Bonsignore M, Barkow K, Jessen F, Heun R. Validity of the five-item WHO Well-Being Index (WHO-5) in an elderly population. Eur Arch Psychiatry Clin Neurosci. 2001;251 Suppl 2:II27-31. doi: 10.1007/BF03035123. PMID 11824831
- [Background] Bech P, Olsen LR, Kjoller M, Rasmussen NK. Measuring well-being rather than the absence of distress symptoms: a comparison of the SF-36 Mental Health subscale and the WHO-Five Well-Being Scale. Int J Methods Psychiatr Res. 2003;12(2):85-91. doi: 10.1002/mpr.145. PMID 12830302
- [Result] Lakes KD, Sharp K, Grant-Beuttler M, Neville R, Haddad F, Sunico R, Ho D, Schneider M, Sawitz S, Paulsen J, Caputo K, Lu KD, Aminian A, Lopez-Ortiz C, Radom-Aizik S. A Six Week Therapeutic Ballet Intervention Improved Gait and Inhibitory Control in Children With Cerebral Palsy-A Pilot Study. Front Public Health. 2019 Jun 25;7:137. doi: 10.3389/fpubh.2019.00137. eCollection 2019. PMID 31294009